CLINICAL TRIAL: NCT02349490
Title: A Multi-centre Proof of Concept Study to Assess Efficacy and Safety of a New Liquid Endoscopic Hemostatic Agent (Seraseal / Fastact ®) in Patients With Active Gastrointestinal Bleeding
Brief Title: Seraseal for Endoscopic Hemostasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Arnulf Ferlitsch, MD, Assoc Prof. PD Dr Arnulf Ferlitsch, Medical University of Vienna
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Seraseal1
Record Dates: First submitted 2015-01-18; First posted 2015-01-29 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Gastrointestinal Hemorrhage
Keywords: gastrointestinal hemorrhage; endoscopy; hemostasis
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A first line therapy (Active Comparator): In group A, Seraseal is applied as initial method for hemostasis. If successful, the bleeding site isthen observed for 5 minutes. If bleeding remains active or recurs the institutional standard of care for hemostasis is applied.
  Interventions: Device: Seraseal / Fastact Hemostatic agent (combined activated factors IIa, VIIa, IXa, Xa )
- Group B rescue therapy (Active Comparator): In group B, Seraseal is applied as rescue therapy after an initial failure of the institutional standard method. If Seraseal was successful, the bleeding site was then observed for 5 minutes. If the bleeding remains active or recurs after Seraseal, alternative methods of hemostasis would be applied.
  Interventions: Device: Seraseal / Fastact Hemostatic agent (combined activated factors IIa, VIIa, IXa, Xa )

INTERVENTIONS:
Device: Seraseal / Fastact Hemostatic agent (combined activated factors IIa, VIIa, IXa, Xa ) — Following endoscopic confirmation of a bleeding, 2,5-5ml of liquid Seraseal / Fastact, is topically applied to the bleeding site via catheter

SUMMARY:
Patients with active gastrointestinal bleeding can be included. 5ml of SerasealTM/Fastact (Wortham Laboratories, Chattanooga, USA), a CE-certified medical product for in human intraoperative use as hemostatic agent, is topically applied via catheters to the bleeding site. In group A, Seraseal is applied as initial method for hemostasis. In group B, Seraseal is applied after an initial failure of the institutional standard method. Homeostatic success is determined by 5 min without bleeding at gastrointestinal site. after application of Seraseal.

DETAILED DESCRIPTION:
Following endoscopic confirmation of a bleeding, 2,5-5ml of liquid Seraseal / Fastact, certified for intraoperative use in humans (CE No 0653), is topically applied to the bleeding site. The delivery device consisted of a 5ml syringe containing Seraseal plugged to standard delivery catheters, either ERCP catheters or dye spraying catheters (Boston Scientific, USA) that are inserted via the working channel of the endoscope. Once the bleeding is identified at endoscopy, the delivery catheter is inserted through the endoscope and positioned toward the lesion, leaving 1-2 cm between the bleeding site and the catheter tip. Seraseal is then delivered in short spray bursts or direct shots (for 1-2 seconds) until hemostasis is confirmed. A maximum of 5ml of Seraseal is administered in each patient. Homeostatic success is determined by 5 min without bleeding at gastrointestinal site. after application of Seraseal.

Two groups are formed for analysis of this proof of concept study:

In group A, Seraseal is applied as initial method for hemostasis. If successful, the bleeding site is then observed for 5 minutes. If bleeding remains active or recurs, the institutional standard of care for hemostasis is applied.

In group B, Seraseal is applied as rescue therapy after an initial failure of the institutional standard method. If Seraseal is successful, the bleeding site is then observed for 5 minutes. If the bleeding remains active or recurs after Seraseal, alternative methods of hemostasis will be applied.

ELIGIBILITY:
Inclusion Criteria:

* active gastrointestinal hemorrhage

Exclusion Criteria:

* no sign of active bleeding at endoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-11; Primary Completion 2013-07 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Hemostasis | 5min
  Success (=Hemostasis) for 5 minutes after Seraseal application

CONTACTS AND LOCATIONS:
Overall Officials: Arnulf Ferlitsch, MD, Principal Investigator — Medical University of Vienna
Locations (4):
- Austria (3):
  - KH der Elisabethinen Linz, Linz, Upper Austria
  - Division of Gastroenterology, Medical University of Vienna, Vienna, Vienna
  - Rudolfstiftung, Vienna, Vienna
- Hannover Medical School, Hanover, Germany

REFERENCES:
- [Derived] Ferlitsch A, Puspok A, Bota S, Wewalka F, Schoefl R, Brownstone E, Madl C, Lenzen H, Lankisch TO, Dolak W, Trauner MH, Ferlitsch M. Efficacy and safety of bovine activated factors IIa/VIIa/IXa/Xa in patients with active gastrointestinal bleeding: a proof of concept study. Endoscopy. 2016 Apr;48(4):380-4. doi: 10.1055/s-0034-1393312. Epub 2015 Nov 12. PMID 26561916